CLINICAL TRIAL: NCT04157842
Title: The Influence of Hip Replacement (Subtrochanteric Osteotomy vs. Non-osteotomy) on Lower Extremity Hemodynamics in Crowe IV Hip Dysplasia Patient
Brief Title: The Influence of Hip Replacement on Lower Extremity Hemodynamics in Crowe IV Hip Dysplasia Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1900025501
Record Dates: First submitted 2019-10-23; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Hip Dysplasia
MeSH Terms: conditions — Hip Dislocation | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total hip replacement with subtrochanteral osteotomy (Experimental): subtrochanteral osteotomy is applied during total hip replacement
  Interventions: Procedure: total hip replacement with subtrochanteral osteotomy
- total hip replacement with no osteotomy (Sham Comparator): no osteotomy is applied during total hip replacement.
  Interventions: Procedure: total hip replacement with no osteotomy

INTERVENTIONS:
Procedure: total hip replacement with subtrochanteral osteotomy — applying subtrochanteral osteotomy during the operation to release the tension of vessels and nerve
  Arms: total hip replacement with subtrochanteral osteotomy
Procedure: total hip replacement with no osteotomy — just total hip replacement
  Arms: total hip replacement with no osteotomy

SUMMARY:
Explore the influence of hip replacement on lower extremity hemodynamics in Crowe Ⅳ hip dysplasia patient.

DETAILED DESCRIPTION:
Changes of limb length after total hip replacement is common, especially for Crowe Ⅳ hip dysplasia patient. Such change potentially increases tension of vessel and influence lower extremity hemodynamics. Till now, little is known in this area.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Crow IV hip dysplasia;
* Bilateral Crow IV hip dysplasia without osteoarthritis on the other side

Exclusion Criteria:

* Patients with serious medical disease;
* Patients with lower extremity vascular disease; 3. Patients with severe mental illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Hip Harris Score | preoperative, 1 week, 6 weeks, 12 weeks, 24 weeks and 1 year after the surgery.
  change of hip harris score scale from baseline(preoperative) to 1 year after surgery.
Leg Length Change | preoperative, 1 week, 6 weeks, 12 weeks, 24 weeks and 1 year after the surgery.
  change of Leg Length from baseline(preoperative) to 1 year after surgery.
Radiographic Results | 1 week, 12 weeks, 24 weeks and 1 year after the surgery.
  change of Radiographic Results from 1 week after surger to 1 year after surgery
Lower Limb Arterial CT Angiography | preoperative, 1 week, 12 weeks after the surgery.
  change of vascular diameter and vascular cross-sectional from baseline(preoperative) to 1 year after surgery baseline(preoperative) to 12 weeks after surgery.
Vascular Ultrasound Examination | preoperative, 1 week, 6 weeks, 12 weeks, 24 weeks and 1 year after the surgery.
  change of systolic peak velocity, end-diastolic velocity, pulsation index, resistance index and blood flow from baseline(preoperative) to 1 year after surgery.
Blood Viscosity | preoperative, 1 week, 6 weeks, 12 weeks, 24 weeks and 1 year after the surgery.
  change of blood viscosity from baseline(preoperative) to 1 year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: SHIGUI YAN, MD, Study Chair — 2nd affiliated hospital, School of Medicine, Zhejiang University